CLINICAL TRIAL: NCT04455113
Title: Hypophosphatemia Deleteriously Affects Outcome of Septic Shock Patients Admitted to ICU
Status: Completed | Type: Observational
Sponsor: Ayman Anis Metry (Other)
Responsible Party: Sponsor-Investigator, Ayman Anis Metry, Assistant professor, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: ASUH612/18
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Effect of Hypophosphatemia on Septic Patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normo-phosphatemia: 238 patients included in this group. Phosphorus level >2.5 mg/dl
  Interventions: Diagnostic Test: Phosphorus level
- Hypophosphatemia: 79 patients included in this group. Phosphorus level <2.5 mg/dl
  Interventions: Diagnostic Test: Phosphorus level

INTERVENTIONS:
Diagnostic Test: Phosphorus level — infusion
  Other Names: sodium-phosphate 10 ml vial

SUMMARY:
Patients with severe sepsis/septic shock complicated by hypophosphatemia are at high risk of developing morbidities other than that underlying sepsis and more vulnerable to higher mortality rate. Thus, the current study hypothesized that diagnosis and management of hypophosphatemia may be advantageous for reduction of morbidity and mortality rates of septic patients admitted to ICU

DETAILED DESCRIPTION:
The current study was started since June 2018 till Jan 2020 after approval of the study protocol by the Local Ethical Committee. The study intended to include all patients admitted to ICU with or developed severe sepsis or septic shock within 24-hr after admission to ICU.

All patients admitted to ICU were eligible to evaluation for demographic and clinical data including hemodynamic data. Disease severity and its impact on body organs were evaluated using acute physiology and chronic health evaluation II score (APACHE II) (20) and SOFA (18) scores. Exclusion criteria included maintenance on immunodepressent therapy for any indication, severe hemorrhagic shock, pregnancy and refusal of nearest relative to sign the written concept for study participation. Children and adulthoods younger than 18 years and patients who were expected to die were also excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to ICU were eligible to evaluation for demographic and clinical data including hemodynamic data.
* Disease severity and its impact on body organs were evaluated using acute physiology and chronic health evaluation II score (APACHE II) (20) and SOFA (18) scores.

Exclusion Criteria:

* Maintenance on immunodepressent therapy.
* Severe hemorrhagic shock.
* Pregnancy
* Refusal of nearest relative to sign the written concept for study participation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included all patients admitted to ICU for sepsis, severe sepsis and septic shock.
  All patients included except mentioned above exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
The 28-day ICU mortality rate (28-MR) | 28 days

SECONDARY OUTCOMES:
The incidence of additional morbidities. | 30 days
The correlation between 28-MR and incidence of additional morbidities and severity of HP. | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No